CLINICAL TRIAL: NCT05311930
Title: Efficacy and Safety of TPO Receptor Agonists as First-line Drugs in the Treatment of Newly Diagnosed Elderly ITP Patients in China-an Open Label Study
Brief Title: Efficacy and Safety of TPO Receptor Agonists in the Treatment of Elderly ITP Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TPO-RAs-old patients
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: hetrombopag; Primary Immune Thrombocytopenia; platelets
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — hetrombopag

STUDY DESIGN:
Intervention Model Description: This is a single-arm open-label trial. After enrollment, patients received an initial dose of 2.5 mg of hetropoda for 4 weeks, and blood routine monitoring was performed regularly during treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2.5mg/d (Experimental): After the subjects signed the informed consent and passed the screening, they entered the treatment period and received a starting dose of 2.5 mg/d of Hetrabopag. During the treatment process, the clinician adjusted the drug dose according to the patient's own conditions. The maximum drug dose was 7.5 mg qd, 28 d Evaluate efficacy and safety after completion;
  Interventions: Drug: 2.5mg/d Hetrombopag

INTERVENTIONS:
Drug: 2.5mg/d Hetrombopag — After the subjects signed the informed consent and passed the screening, they entered the treatment period and received a starting dose of 2.5 mg/d of Hytrombopag. During the treatment process, the clinician adjusted the drug dose according to the patient's own conditions. The maximum drug dose was 7.5 mg qd, 28 d Evaluate efficacy and safety after completion;
  Other Names: no use

SUMMARY:
Elderly ITP patients have many underlying diseases, hormone contraindications and many adverse reactions during the use of hormones. TPO-RAs are oral small-molecule non-peptide drugs. Retrospective studies have shown that they have good efficacy and high safety in elderly patients. Therefore, this study is a prospective trial to evaluate TPO-RAs as the first-choice drug for the treatment of elderly ITP patients with contraindications to hormones, aiming to improve the efficacy-risk ratio of elderly patients

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an immune disorder characterized by decreased production and increased destruction of platelets. In recent years, with the in-depth exploration of its pathogenesis and the continuous influx of new drugs, the status of second-line treatment drugs, mainly TPO receptor agonists (TPO-RAs), has been continuously improved, which has brought great importance to the treatment and management of ITP patients. However, for elderly ITP patients with severe underlying diseases, poor hormone tolerance, severe adverse reactions or hormone contraindications, whether TPO receptor agonists can be used as the first-choice drug and its efficacy and safety are still lacking relevant research, and for elderly ITP patients There is a lack of uniform guidelines for the treatment and management of patients. Limited retrospective studies have shown that TPO receptor agonists have good safety and efficacy, and are expected to become the recommended drugs for the treatment of elderly patients with ITP. However, whether TPO receptor agonists can be directly used as the first-choice drug for newly diagnosed elderly ITP patients who are not suitable for first-line treatment and its efficacy are uncertain.

This study will include newly diagnosed elderly ITP patients with hormonal contraindications or potential serious side effects of hormonal therapy, take the TPO-RA drug hetropoda as the first-choice treatment drug, and explore the effectiveness of hetrompopag in such patients and safety analysis. This study will provide new ideas and clinical basis for standardized and individualized treatment of elderly ITP patients, and provide practical experience for promoting the establishment of elderly ITP treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient voluntarily signed the informed consent; 2. The patient is a newly diagnosed ITP patient, aged ≥60 years old; 3. Two consecutive PLTs < 30×109/L, or two consecutive PLTs < 30×109/L≤PLT<50×109/L but with risk factors such as bleeding (such as previous bleeding history and/or anticoagulation/antiplatelet) Concomitant medication) or age > 75 years; 4. Have not received first-line treatment such as hormones, IVIG, etc.; 5. There is any hormonal contraindication (with active peptic ulcer, recent gastrointestinal anastomosis, corneal ulcer, severe hypertension (high blood pressure ≥ grade 2), diabetes with poor blood sugar control, infection that cannot be controlled by antibiotics ( Bacterial and viral infections), heart failure and adrenal hyperfunction, severe mental illnesses such as epilepsy, severe osteoporosis, rheumatoid arthritis, tuberculosis, fractures, patients with combined antithrombotic and antiplatelet drugs, etc.); 6. The following clinical biochemical indicators must be within ±20% of the upper and lower limits of normal values: creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin and alkaline phosphatase.

Exclusion Criteria:

* 1. Exclude immune diseases such as systemic lupus erythematosus, antiphospholipid syndrome, etc.; 2. Exclude drug-related thrombocytopenia; 3. Bone marrow-related examinations suggest the presence of other primary diseases of the blood system (such as MDS, AA, thrombotic thrombocytopenic purpura, etc.) or the presence of myelofibrosis MF≥2; 4. Participated in other clinical trials affecting platelet count and function 3 months before the trial; 5. Previously received first-line therapy such as hormones, IVIG; 6. Previous use of TPO-RAs or poor efficacy against known TPO drugs; 7. The patient has experienced severe arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), or clinical symptoms suggest thrombophilia; 8. HIV, hepatitis B or C seropositive or a history of liver cirrhosis or portal hypertension; 9. Life-threatening bleeding (WHO bleeding score 4) or the patient is expected to require salvage treatment before the first dose; 10. Has a history of malignant tumor or is accompanied by malignant tumor; 11. The investigator believes that there are any other circumstances that may cause the subjects to fail to complete the study or bring obvious risks to the subjects.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 28 days
  Proportion of subjects with platelet counts ≥50×10^9/L after 28 days of treatment

SECONDARY OUTCOMES:
Remission rate | 28 days
  Complete response, effective, ineffective proportion of testers after 28 days of treatment
Drug efficacy | 28 days
  During treatment, the proportion of subjects, which the platelet count at least once reached ≥50×109/L.
Evaluation of effectiveness | 28 days
  During treatment, the proportion of subjects, which the platelet count increased at least 2 times compared with baseline.
Adverse events | 6 months from treatment
  Evaluate the incidence and severity of bleeding based on the ITP-BAT bleeding score
Adverse events | 6 months from treatment
  During treatment, the proportion of subjects, which received at least once rescue
Side effects of drugs | 1 month from treatment
  Assessing safety through the adverse events,such as liver damage, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
the data will share to others if they not involve patient privacy
Supporting Information: Study Protocol
Time Frame: the data will be shared after the study is completed, it will take 2 years.
Access Criteria: Not sure yet

REFERENCES:
- [Background] Frederiksen H, Schmidt K. The incidence of idiopathic thrombocytopenic purpura in adults increases with age. Blood. 1999 Aug 1;94(3):909-13. PMID 10419881
- [Background] Moulis G, Palmaro A, Montastruc JL, Godeau B, Lapeyre-Mestre M, Sailler L. Epidemiology of incident immune thrombocytopenia: a nationwide population-based study in France. Blood. 2014 Nov 20;124(22):3308-15. doi: 10.1182/blood-2014-05-578336. Epub 2014 Oct 10. PMID 25305203
- [Background] Glynn RJ, Field TS, Rosner B, Hebert PR, Taylor JO, Hennekens CH. Evidence for a positive linear relation between blood pressure and mortality in elderly people. Lancet. 1995 Apr 1;345(8953):825-9. doi: 10.1016/s0140-6736(95)92964-9. PMID 7898229
- [Background] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Background] Cortelazzo S, Finazzi G, Buelli M, Molteni A, Viero P, Barbui T. High risk of severe bleeding in aged patients with chronic idiopathic thrombocytopenic purpura. Blood. 1991 Jan 1;77(1):31-3. PMID 1984800
- [Background] Ruggeri M, Tosetto A, Palandri F, Polverelli N, Mazzucconi MG, Santoro C, Gaidano G, Lunghi M, Zaja F, De Stefano V, Sartori R, Fazi P, Rodeghiero F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Anemia and Thrombocytopenias Working Party. GIMEMA Study ITP0311. Thrombotic risk in patients with primary immune thrombocytopenia is only mildly increased and explained by personal and treatment-related risk factors. J Thromb Haemost. 2014 Aug;12(8):1266-73. doi: 10.1111/jth.12636. Epub 2014 Jul 16. PMID 24942752
- [Background] Michel M, Rauzy OB, Thoraval FR, Languille L, Khellaf M, Bierling P, Godeau B. Characteristics and outcome of immune thrombocytopenia in elderly: results from a single center case-controlled study. Am J Hematol. 2011 Dec;86(12):980-4. doi: 10.1002/ajh.22170. Epub 2011 Sep 28. PMID 21956157
- [Background] Daou S, Federici L, Zimmer J, Maloisel F, Serraj K, Andres E. Idiopathic thrombocytopenic purpura in elderly patients: a study of 47 cases from a single reference center. Eur J Intern Med. 2008 Oct;19(6):447-51. doi: 10.1016/j.ejim.2007.07.006. Epub 2008 Feb 20. PMID 18848179
- [Background] Zhou H, Fu R, Wang H, Zhou F, Li H, Zhou Z, Zhang L, Yang R. Immune thrombocytopenia in the elderly: clinical course in 525 patients from a single center in China. Ann Hematol. 2013 Jan;92(1):79-87. doi: 10.1007/s00277-012-1567-2. Epub 2012 Sep 6. PMID 22956151